CLINICAL TRIAL: NCT04967534
Title: The Efficacy of Whole-Body Electromyostimulation (WB-EMS) in Frail Older People: A Randomized Controlled Trial
Brief Title: Efficacy of WB-EMS in Frail Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETAPPEN_MAIN
Record Dates: First submitted 2021-07-15; First posted 2021-07-19 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2021-07

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: parallel-group (1:1) randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WB-EMS (Experimental)
  Interventions: Behavioral: WB-EMS
- social contact control group (Sham Comparator)
  Interventions: Behavioral: social contact control group

INTERVENTIONS:
Behavioral: WB-EMS — Simultaneous, individually adjustable stimulation of 12 muscle groups using an interval approach with a duty cycle of 6s impulse/4s rest, bipolar electric current (impulse -frequency 85Hz, -width 350μs, rectangular pattern) will be applied. After a 4-week conditioning period, 1.5x 20 min/week WB-EMS will be conducted for 12 weeks (total training duration 8 weeks). Easy to perform functional exercises focusing on balance, transfer ability, stepping, and lower extremity strength will be done during WB-EMS. Exercise intensity will be individually prescribed and adjusted by the rate of perceived exertion (RPE-Borg CR10 scale 4 (moderate) to 7 (hard)). WB-EMS will be fully supervised one-on-one.
  Arms: WB-EMS
Behavioral: social contact control group — Psycho-social intervention with participants randomized to the control group receiving (if wanted) the same social contact time (20-30 minutes/week) as the WB-EMS group. Depending on personal preferences and Covid-19 restrictions this will be done by phone or in-person one-on-one. Health-related topics and/or general chatting will be offered.
  Arms: social contact control group

SUMMARY:
Exercise in general and resistance training (RT) in particular have demonstrated positive effects on frailty outcomes, including physical functioning. However, frail older people with functional impairments are among the least physically active and have problems reaching high-intensity levels. Whole-body electromyostimulation (WB-EMS) allows the simultaneous innervation of all large muscle groups by external electrical stimulation, inducing a high-intensity RT at a low subjective effort level. The efficacy of WB-EMS in frail older people has yet to be determined.

The primary objective of this study is to investigate the efficacy of WB-EMS in frail older people.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years and older
* frail according to Tilburg Frailty Indicator
* residing in assisted living facility or nursing home
* able to walk 4m w/o walking aid but without personal assistance
* no prior WB-EMS exposure

Exclusion Criteria:

* severe visual or hearing impairments
* major cognitive impairment (MMSE <10)
* medications with muscle-anabolic effects
* medical conditions affecting trainability of muscles (e.g. Myasthenia gravis, Cushing syndrome, Morbus McArdle)
* surgery within past two months
* history of rhabdomyolysis
* medical conditions affecting sensation of electrical stimuli (e.g. severe polyneuropathy)
* severe renal insufficiency (eGFR<30 ml/min/1.73m²)
* electronic implants
* acute or untreated abdominal wall or inguinal hernia
* Ventricular arrhythmias requiring therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Lower Extremity Functioning | 8 weeks, 16 weeks, 32 weeks
  The Short Physical Performance Battery (SPPB) comprises of three dimensions, balance (static - standing in 3 positions of increasing difficulty by reducing base of support for max. 10s), gait (usual pace - two walks of 4m lengths), functional strength (chair rise - five times sit-to-stand transfers as fast as possible). A sum score is calculated (0-12 points) with higher scores indicating better functional status and each dimension being equally weighed (0-4 points).

SECONDARY OUTCOMES:
Change in Mobility measured by the Timed up & go test (TUG) | 8 weeks, 16 weeks, 32 weeks
  The TUG requires the participants to stand up from a chair, walk at usual pace to line at 3m, turn, walk back and sit down again. The time in seconds is recorded.
Change in leg strength | 8 weeks, 16 weeks, 32 weeks
  Maximal isometric knee extension strength will be assessed on the dominant leg with the participant seated. Three trials will be conducted.
Change in maximal hand grip strength | 8 weeks, 16 weeks, 32 weeks
  Grip strength will be assessed on the dominant hand using a digital dynamometer with the participant seated. Three trials will be conducted.
Change in gait speed | 16 weeks, 32 weeks
  Gait speed will be assessed over 6 meters under 3 conditions, 1) walking at usual pace, 2) walking at usual pace while counting backwards by 3, 3) walking at fast pace
Change in Choice Stepping Reaction Time (CSRT) test | 16 weeks, 32 weeks
  CSRT time will be measured as the total time to complete 12 steps onto four targets printed on a portable rubber mat following 8 practice trials.
Change in Body Sway | 8 weeks, 16 weeks, 32 weeks
  An instrumented test of postural sway (ISway) using a body-worn accelerometer will be used.
Change in Balance performance | 16 weeks, 32 weeks
  The Berg Balance Scale (BBS) will be used to assess 14 balance tasks of static and dynamic stability. Each task is scored on a five-point scale according to quality or time ranging from "0" (lowest level of function) to "4" (highest level). The maximum score is 56.
Change in Functional Balance | 16 weeks, 32 weeks
  The Alternate Step Test (AST) measures the time required to place the feet eight times in alternate order on a sturdy step (18 cm high) as fast as possible
Change in Frailty Status | 16 weeks, 32 weeks
  Frailty will be assessed by the Fried Phenotype and the Tilburg Frailty Indicator (TFI).
  The Fried phenotype comprises of muscle weakness, fatigue, slowness, low physical activity levels, unintentional weight loss, each scored as 0 (criterion not fulfilled) or 1 (criterion fulfilled). A total sum score of 0 indicates a person is robust, a score of 1 or 2 indicates pre-frailty and a score of 3-5 indicates frailty.
  The TFI is a self-reported frailty scale consisting of 3 domains, physical (8 items), psychological (4 items) and social (3 items). A total sum score greater or equal to 5 indicates frailty.
Change in lean mass | 16 weeks, 32 weeks
  Lean mass will be assessed using Bioelectrical Impedance Analysis (BIA).
Change in fat mass | 16 weeks, 32 weeks
  Fat mass will be assessed using Bioelectrical Impedance Analysis (BIA).
Change in Physical Activity | 16 weeks
  Physical activities will be assessed using a 7-day accelerometry measurement. The device (ActivPAL 3 micro) will be attached to participants' thigh and worn over the complete 7-day/24-hour period.
Change in concentration of Triglycerides | 16 weeks
  Concentration of Triglycerides measured in mg/dl before first and last trainings
Change in concentration of total cholesterol | 16 weeks
  Concentration of Cholesterin measured in mg/dl before first and last trainings
Change in concentration of high-density lipoprotein (HDL) | 16 weeks
  Concentration of HDL measured in mg/dl before first and last trainings
Change in concentration of low-density lipoprotein (LDL) | 16 weeks
  Concentration of LDL measured in mg/dl before first and last trainings
Change in concentration of glucose | 16 weeks
  Concentration of Glucose measured in mg/dl before first and last trainings
Change in concentration of Creatinkinase (CK) | 8 weeks, 16 weeks
  Concentration of CK measured in U/l before the first and after the last training
Change in concentration of Creatinine | 8 weeks, 16 weeks
  Concentration of Creatinine measured in mg/dl before the first and after the last training
Change in estimated glomerular filtration rate (eGFR) | 8 weeks, 16 weeks
  eGFR (creatinine clearance) measured in mL/min/1.73m² before the first and after the last training
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 8 weeks, 16 weeks
  Pain and function due to orthopedic problems will be assessed with the WOMAC questionnaire, comprising of 24 items each scored on a 5-point Likert scale.
Change in continence status | 16 weeks, 32 weeks
  Continence status (frequency, severity, perceived burden, timing) will be assessed using the International Consultation on Incontinence Questionnaire (ICIQ, 5 items) and the short form of the Urogenital Distress Inventory (UDI-6, 6 items).
Change in depressive symptoms | 16 weeks, 32 weeks
  Depressive symptoms will be assessed using the Iowa version of the Center for Epidemiologic Studies Depression Scale (CES-D), consisting of 11 items, each scored on a 3-point rating scale. The total sum score is calculated.
Change in concerns about falling | 16 weeks, 32 weeks
  The Falls-efficacy Scale-International (FES-I) questionnaire will be used to assess the concerns about falling during 16 activities of daily living. Each item is scored on a 4-point rating scale and the total sum score is calculated.
Change in Quality of Life (QoL) | 16 weeks
  QoL will be assessed with 26-item WHOQOL-BREF covering physical health, psychological health, social relationships and environmental aspects. Each item is scored on a 5-point Likert scale.
Change in sarcopenia specific QoL | 16 weeks, 32 weeks
  Sarcopenia specific QoL will be assessed with the SarQoL, comprising of 55 items in 22 questions rated on a 4-point Likert scale. Seven domains are specified: Physical and mental health, Locomotion, Body composition, Functionality, Activities of daily living, Leisure activities and Fear.
Change in Health-related Quality of Life (HrQoL) | 8 weeks, 16 weeks, 32 weeks
  HrQoL will be assessed using the 4-item HowRu scale comprising of 4 variables: pain or discomfort, feeling low or worried, limitation in activities and dependency on others. Each item is scored on a 4-point visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kemmler, PhD, Principal Investigator — University of Erlangen-Nürnberg Medical School
Locations (1):
- Institute of Medical Physics, University of Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request by the principal investigator. IPD relevant to a specific publication will be shared deidentified if it is the respective journal's requirement.
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to wolfgang.kemmler@imp.uni-erlangen.de